CLINICAL TRIAL: NCT06376227
Title: With or Without Left Colic Artery Preservation
Brief Title: Robotic-Assisted or Laparoscopic Radical Resection for Rectal Cancer With or Without Left Colic Artery Preservation
Status: Completed | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Daorong Wang, Doctor, Northern Jiangsu People's Hospital
Other Study IDs: jamesdukeryan
Record Dates: First submitted 2024-04-10; First posted 2024-04-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Rectal Cancer; Left Colic Artery Stenosis (Diagnosis); Robotic Assisted Laparoscopic Surgery
Keywords: Rectal cancer; Left colic artery; High ligation; Low ligation; Inferior mesenteric artery; Robotic-assisted laparoscopy
MeSH Terms: conditions — Rectal Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with or without Left Colic Artery Preservation
- low ligation (LL) group and high ligation (HL) group: low ligation (LL) which with preservation of LCA and high ligation (HL) which without preservation of LCA
  Interventions: Procedure: with or without Left Colic Artery Preservation

INTERVENTIONS:
Procedure: with or without Left Colic Artery Preservation — low ligation (LL) which with preservation of LCA and high ligation (HL) which without preservation of LCA
  Groups: low ligation (LL) group and high ligation (HL) group

SUMMARY:
Brief Summary

Background The preservation of the left colic artery (LCA) during rectal cancer resection remains a topic of controversy, and there is a notable absence of robust evidence regarding the outcomes associated with LCA preservation. And the advantages of robotic-assisted laparoscopy (RAL) surgery in rectal resection remain uncertain. The objective of this study was to assess the influence of LCA preservation surgery and RAL surgery on intraoperative and postoperative complications of rectal cancer resection.

Methods Participants who underwent laparoscopic (LSC) or RAL with or without LCA preservation resection for rectal cancer between April 2020 and May 2023 were retrospectively assessed. The patients were categorized into two groups: low ligation (LL) which with preservation of LCA and high ligation (HL) which without preservation of LCA. A one-to-one propensity score-matched analysis was performed to decrease confounding. The primary outcome was operative findings, operative morbidity, and postoperative genitourinary function.

DETAILED DESCRIPTION:
The investigators retrospectively collected data from the medical records of participants who had rectal cancer at Northern Jiangsu People's Hospital, from April 2020 to May 2023. A total of 612 from 1164 cases were included in this study; in 462 cases, the LCA was preserved by LL intraoperatively (LL group), in which 202 cases underwent robotic-assisted laparoscopy (LL-RAL subgroup) and 260 cases underwent laparoscopy (LL-LSC subgroup). While in the remaining 150 cases, the LCA was not preserved by HL intraoperatively (HL group). in which 70 cases underwent robotic-assisted laparoscopy (HL-RAL subgroup) and 80 cases underwent laparoscopy (HL-LSC subgroup).

ELIGIBILITY:
Inclusion Criteria:

* Low anterior resection for rectal cancer
* Postoperative pathological diagnosis of rectal adenocarcinoma
* Informed consent signed prior to surgery.

Exclusion Criteria:

* Recurrent rectal cancer
* Emergency surgery
* Preoperative and intraoperative detection of distant organ metastases or extensive
* Implantation metastases in the abdominal cavity
* Palliative surgery
* A postoperative pathology report that showed residual cancer cells at the proximal or distal resection margin
* No standard chemotherapy for tumor-node-metastasis (TNM) staging II or III after surgery
* Synchronous colorectal carcinoma and other organ tumors
* Incomplete case data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 612 rectal cancer patients, including 245 (40.0%) men and 367(60.0%) women, were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1164 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
The incidence of anastomotic leakage in postoperative patients with or without left colic artery preservation. | 2 weeks within the surgery
  Within two weeks after surgery, the patient experienced abdominal pain, fever, and imaging diagnosis showed anastomotic leakage.

SECONDARY OUTCOMES:
The genitourinary function of the patients after the radical resection with or without left colic artery preservation. | 6 to 12 months after operation
  The genitourinary function includes urinary dysfunction and sexual dysfunction. Residual urine volume and catheterization retention time for evaluating urinary function. Erectile and ejaculatory grading scores are used to evaluate sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Daorong Wang, M.D., Professor, Study Director — Northern Jiangsu People's Hospital
Locations (1):
- Northern Jiangsu People's Hospital Affiliated to Yangzhou University, General Surgery Institute of Yangzhou, Yangzhou University , Yangzhou, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Contains a large amount of personal information about patients and needs to be treated with caution.